CLINICAL TRIAL: NCT01124058
Title: Evaluation of Maintenance Dosing vs Loading Dosing Upon Restarting Warfarin Therapy: A Prospective Randomized Trial.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Tammy Bungard, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007UHFMDvsLD
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Anticoagulation
Keywords: restarting warfarin; time to therapeutic INR
MeSH Terms: interventions — Warfarin; Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loading (Experimental): 1.5 times the maintenance dose for 3 days, then resumption of warfarin dosing as per the maintenance dose
  Interventions: Drug: warfarin
- Maintenance (Active Comparator): Re-start same dose as previously stable on
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: warfarin — Patients will be randomized to re-start warfarin at their "maintenance" dose or at a "loading" dose (1.5 times the maintenance dose for 3 days, then resumption of warfarin dosing as per the maintenance dose).
  Other Names: warfarin, Taro-warfarin, Apo-warfarin, Coumadin, Fragmin, Low-molecular weight heparin
  Arms: Loading
Drug: Warfarin — "Maintenance" dose is the amount of warfarin that a patient required to maintain a therapeutic INR.
  Other Names: warfarin, Taro-warfarin, Apo-warfarin, Coumadin, Fragmin, Low-molecular weight heparin
  Arms: Maintenance

SUMMARY:
A prospective, randomized trial to compare the time taken to achieve a therapeutic INR upon re-starting warfarin at a "loading" dose (namely 1.5 times the "maintenance" dose for 3 days) compared to the known "maintenance" dose.

DETAILED DESCRIPTION:
Patients will be identified via the University of Alberta Hospital Anticoagulation Management Service. Following the receipt of written, informed consent, patients will be randomized to re-start warfarin at their "maintenance" dose or at a "loading" dose (1.5 times the maintenance dose for 3 days, then resumption of warfarin dosing as per the maintenance dose). Randomization will be performed on-line through the EPICORE Centre.

Assuming Day 1 is the day warfarin is re-started, patients will have INRs done on day 3 and at least every 2 days thereafter until a therapeutic INR is obtained. In addition, protein C, protein S and factor II levels will be obtained while the patient is on stable maintenance dosing of warfarin (i.e., prior to holding warfarin for the procedure), 7 days after re-starting warfarin, and 14 days after re-starting warfarin. Complete blood counts (CBCs) will be done with each INR if the patient is taking a low molecular weight heparin (LMWH). Patients will have their anticoagulant therapy managed by the AMS for 6 weeks and will receive a telephone follow-up by the AMS at 90 days to determine if any bleeding or clotting complications occurred.

ELIGIBILITY:
Inclusion Criteria:

* Have 'stable warfarin maintenance dosing' (defined as last 2 INRs within therapeutic range with weekly warfarin dosing not being changed any more than 10%)
* Have an INR indicative of not taking any warfarin (INR <1.4) or confirmation of the patient not taking any warfarin in the past 4 days
* Provide written, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
re-starting warfarin "loading" dose vs "maintenance" dose | INR drawn 3 days post-reinitiation and then every 2 days until therapeutic
  To compare the time taken to achieve a therapeutic INR between those patients re-starting warfarin with a "loading" dose and a "maintenance" dosing regimen using linear interpolation of INRs.

SECONDARY OUTCOMES:
Compare % of time within, above and below the target INR range | days
  To compare the % of time within, above and below the desired INR range between those patients re-starting warfarin with a "loading" dose or "maintenance" dose 6 weeks following restarting warfarin.
Compare bleeding/clotting complications between two groups | 30 days, 90 days
  To compare the rates of thrombosis (i.e., stroke) / major hemorrhage between those re-starting warfarin with a "loading" dose or "maintenance" dose at 30 days and 90 days following restarting warfarin.
Compare the levels of protein C, protein S, and factor II between 2 groups. | week
  To compare the levels of protein C, protein S, and factor II between those re-starting warfarin with a "loading" dose or "maintenance" dose.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy J Bungard, BSP, PharmD, Principal Investigator — Univeristy of Alberta; Bruce Ritchie, MD, FRCPC, Principal Investigator — University of Alberta
Locations (1):
- Univeristy of Alberta, Edmonton, Alberta, Canada